CLINICAL TRIAL: NCT07269392
Title: Impact of Dual Trigger Using Recombinant Human Chorionic Gonadotropin (HCG) and Gonadotropin-releasing Hormone (GnRH) Agonist on Thawed Modified Natural Cycle Outcomes: an Open-label Multi-center Randomized Controlled Trial.
Brief Title: Dual Trigger With HCG and GnRH Agonist on Thawed Modified Natural Cycle Embryo Transfer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202409081MINB
Record Dates: First submitted 2025-09-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: In Vitro Fertilization (IVF); Embryo Transfer
MeSH Terms: interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dual (Experimental): GnRH agonist
  Interventions: Drug: GnRH agonist
- hcg (No Intervention): hcg

INTERVENTIONS:
Drug: GnRH agonist — GnRH agonist add to hcg for trigger
  Arms: dual

SUMMARY:
Impact of dual trigger using recombinant human chorionic gonadotropin (HCG) and gonadotropin-releasing hormone (GnRH) agonist on thawed modified natural cycle outcomes: an open-label multi-center randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. 24<= Age < 45 patient undergo mNC-FET

Exclusion Criteria:

1. Congenital or acquired uterine abnormalities (uterine malformation, submucosal myoma, intrauterine adhesion or endometrial polyp >1cm)

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Implantation | 14 days after embryo transfer
  Implantation is defined as a positive serum β-hCG (>20 mIU/mL) measured 14 days after embryo transfer.

SECONDARY OUTCOMES:
Clinical pregnancy | one week after confirm pregnancy
  Clinical pregnancy is defined as visualization of a gestational sac on transvaginal ultrasonography one week after pregnancy has been confirmed.
Ongoing pregnancy rate | 5 weeks after confirmed pregnancy
  An ongoing pregnancy is defined as a viable intrauterine pregnancy with fetal cardiac activity at ≥9 weeks' gestational age.
Miscarriage rate | before delivery
Gestational age (weeks) at delivery | delivery
  Gestational age (weeks) at delivery
Live birth rate | delivery
Birth weight | delivery
  Birth weight of the bewborn (kg)
Presence of significant congenital or medical conditions of the newborn | delivery
  Presence of significant congenital or medical conditions of the newborn

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haas J, Bassil R, Samara N, Zilberberg E, Mehta C, Orvieto R, Casper RF. GnRH agonist and hCG (dual trigger) versus hCG trigger for final follicular maturation: a double-blinded, randomized controlled study. Hum Reprod. 2020 Jul 1;35(7):1648-1654. doi: 10.1093/humrep/deaa107. PMID 32563188
- [Background] Lin MH, Wu FS, Hwu YM, Lee RK, Li RS, Li SH. Dual trigger with gonadotropin releasing hormone agonist and human chorionic gonadotropin significantly improves live birth rate for women with diminished ovarian reserve. Reprod Biol Endocrinol. 2019 Jan 4;17(1):7. doi: 10.1186/s12958-018-0451-x. PMID 30609935
- [Background] Wang Y, Yi YC, Guu HF, Chen YF, Kung HF, Chang JC, Chen LY, Chuan ST, Chen MJ. GnRH agonist-only trigger, compared to dual trigger, reduces oocyte retrieval rate in high responders without affecting cumulative live birth rate. Front Endocrinol (Lausanne). 2024 Aug 20;15:1461317. doi: 10.3389/fendo.2024.1461317. eCollection 2024. PMID 39229374
- [Background] Halim B, Lubis HP. Dual trigger with gonadotropin-releasing hormone agonist and recombinant human chorionic gonadotropin improves the outcome of intrauterine insemination. Obstet Gynecol Sci. 2022 Mar;65(2):207-214. doi: 10.5468/ogs.21275. Epub 2022 Feb 21. PMID 35184525
- [Background] Yildirim Kopuk S, Ece Utkan Korun Z, Yuceturk A, Karaosmanoglu O, Yazicioglu C, Tiras B, Cakiroglu Y. Does dual trigger improve euploidy rate in normoresponder? A cross-sectional study. Int J Reprod Biomed. 2023 May 12;21(5):395-402. doi: 10.18502/ijrm.v21i5.13473. eCollection 2023 May. PMID 37362090
- [Background] He Z, Liu Y, Huang N, Liu X, Zeng L, Lian Y, Li R, Chi H. Dual trigger versus human chorionic gonadotropin trigger for blastocyst quality and cumulative live birth. J Assist Reprod Genet. 2024 Dec;41(12):3445-3453. doi: 10.1007/s10815-024-03293-5. Epub 2024 Nov 16. PMID 39549203
- [Background] Hu KL, Wang S, Ye X, Zhang D, Hunt S. GnRH agonist and hCG (dual trigger) versus hCG trigger for follicular maturation: a systematic review and meta-analysis of randomized trials. Reprod Biol Endocrinol. 2021 Jun 1;19(1):78. doi: 10.1186/s12958-021-00766-5. PMID 34059045